CLINICAL TRIAL: NCT06547164
Title: A Phase I, Open-label, 2 Part, Fixed Sequence Study to Assess the Effect of Co-administration of Camizestrant (AZD9833) on the Pharmacokinetics of Midazolam Exposure (CYP3A4/5 Substrate) and of Carbamazepine (CYP3A4/5 Inducer) on Camizestrant Exposure in Healthy Post Menopausal Female Participants
Brief Title: A Study to Investigate the Pharmacokinetics of Midazolam After Repeated Doses of Camizestrant (AZD9833) and to Investigate the Pharmacokinetics of Camizestrant When Administered Alone and in Combination With Carbamazepine in Healthy Post-Menopausal Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8532C00006
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: Midazolam; Camizestrant; Carbamazepine; Post-menopausal; Estrogen receptor (ER) positive disease; Breast Cancer; Cytochrome P450, family 3, subfamily A (CYP3A)
MeSH Terms: conditions — Breast Neoplasms | interventions — Midazolam; AZD9833; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: Midazolam + Camizestrant (Experimental): Participants will receive a single oral dose of midazolam on Day 1 in Period 1, followed by oral dose of camizestrant OD from Day 2 to Day 6 in Period 2, and then single oral dose of midazolam with camizestrant on Day 7 with PK sampling on Day 7 to Day 8 in Period 3.
  Interventions: Drug: Midazolam; Drug: Camizestrant
- Part B: Camizestrant + Carbamazepine (Experimental): Participants will receive a single oral dose of camizestrant on Day 1 with PK sampling on Day 1 to Day 4 in Period 1, followed by low oral doses of carbamazepine BID on Day 4 to Day 6, mid oral doses of carbamazepine BID on Day 7 to Day 9 and high oral doses of carbamazepine BID on Day 10 to Day 15 with single oral dose of camizestrant on Day 13 with PK sampling on Day 16 in Period 2.
  Interventions: Drug: Camizestrant; Drug: Carbamazepine

INTERVENTIONS:
Drug: Midazolam — Midazolam will be administered orally.
  Arms: Part A: Midazolam + Camizestrant
Drug: Camizestrant — Camizestrant will be administered orally.
  Other Names: AZD9833
Drug: Carbamazepine — Carbamazepine will be administered orally.
  Arms: Part B: Camizestrant + Carbamazepine

SUMMARY:
This study will be conducted in order to determine the effect of repeated oral doses of camizestrant on the pharmacokinetics (PK) of midazolam and to determine the effect of repeated oral titrated doses of carbamazepine on the PK of camizestrant in healthy post-menopausal female participants.

DETAILED DESCRIPTION:
This is an open-label, fixed sequence, 2-part (Part A and Part B), drug-drug interaction study in healthy post-menopausal female participants. Participants enrolled in Part A may subsequently also participate in Part B.

Part A of the study will assess the effect of repeated oral doses of camizestrant on the PK of a single oral dose of midazolam. It will comprise:

* A Screening Period of maximum 28 days.
* Three Treatment Periods during which participants will be resident at the Clinical Unit from the day before study intervention administration (Day -1) until after the last camizestrant PK sample on Day 8.

  1. Period 1: participants will receive a single oral dose of midazolam (Day 1).
  2. Period 2: participants will receive an oral once daily (OD) dose of camizestrant (Day 2 to Day 6).
  3. Period 3: participants will receive a single oral dose of midazolam and camizestrant (Day 7).
* A Follow-up Visit, for which the participant will return to the Clinical Unit 7 (± 2) days after the last camizestrant PK sample in Period 3.

Part B of the study will assess the effect of multiple oral doses of carbamazepine on the PK of a single oral dose of camizestrant. It will comprise:

* A Screening Period of maximum 28 days.
* Two Treatment Periods during which participants will be resident at the Clinical Unit from the day before study intervention administration (Day -1) until after the last camizestrant PK sample on Day 16.

  1. Period 1: participants will receive a single oral dose of camizestrant (Day 1) with PK sampling on Day 1 to Day 4.
  2. Period 2: participants will receive low oral doses (Dose 1) of carbamazepine twice a day (BID) on Day 4 to Day 6, mid oral doses (Dose 2) of carbamazepine BID on Day 7 to Day 9, and high oral doses (Dose 3) of carbamazepine BID on Day 10 to Day 15. On Day 13, participants will receive a single oral dose of camizestrant.
* A Follow-up Visit, for which the participant will return to the Clinical Unit 7 (± 2) days after the last camizestrant PK sample in Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy post-menopausal female participants with suitable veins for cannulation or repeated venipuncture.
* Female participants must be post-menopausal as confirmed at the Screening Visit. Post-menopausal defined as amenorrhoea for at least 12 months or more without an alternative medical or surgical cause and confirmed by a follicle stimulating hormone (FSH) result of ≥ 30 Internation units/liter (IU/L).
* Have a body mass index between 19 and 35 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
* Must agree to not use warfarin or phenytoin (and other coumarin-derived vitamin K antagonist anticoagulants) during the study, and for 2 weeks after last administration of study intervention.

Exclusion Criteria:

* History of any clinically important disease or disorder.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of any clinically significant cardiovascular, chronic respiratory disease, haematological, neurological or psychiatric disorder.
* History of acute pulmonary insufficiency marked neuromuscular respiratory weakness, obsessional states, phobic states, sleep apnoea syndrome, and unstable myasthenia gravis.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Any clinically important abnormalities in clinical chemistry, haematology, or urinalysis results.
* Any relevant history or known risk factors of QT prolongation or have received drugs known to prolong QT interval.
* Any positive result for serum Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV).
* History of or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to camizestrant or the formulation excipients.
* Presence of any contraindication to the probe substrate carbamazepine.
* Presence of any contraindication to midazolam.
* Have any active indication for therapeutic anticoagulation, and/or having taken an anticoagulant within 14 days of Screening Visit.
* Part B only: Participants identified to carry human leukocyte antigen (HLA)-A*3101 and/or HLA-B*1502 allele.
* Participants with bone marrow suppression or a history of bone marrow suppression or aplastic anaemia.
* History of or ongoing clinically significant visual disturbances including but not limited to visual hallucinations, migraine with visual symptoms, blurred vision, frequent floaters/flashes associated with other symptoms such as dizziness.
* Participants with family history of glaucoma or closed angle glaucoma or participants who are currently on anticholinergic medications.
* Participants with an anticipated need for major surgery and/or any surgery requiring general anaesthesia during the participation in the study.
* Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy post-menopausal female
Enrollment: 40 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Part A: Area under concentration-time curve from time 0 to infinity (AUCinf) of midazolam | Period 1 (Day 1) and Period 3 (Day 7 to Day 8)
  To determine the effect of repeated oral doses of camizestrant on the key PK parameters of a single oral dose of midazolam in healthy postmenopausal female participants.
Part A: Area under concentrationcurve from time 0 to the last quantifiable concentration (AUClast) of midazolam | Period 1 (Day 1) and Period 3 (Day 7 to Day 8)
  To determine the effect of repeated oral doses of camizestrant on the key PK parameters of a single oral dose of midazolam in healthy postmenopausal female participants.
Part A: Maximum observed plasma (peak) drug concentration (Cmax) of midazolam | Period 1 (Day 1) and Period 3 (Day 7 to Day 8)
  To determine the effect of repeated oral doses of camizestrant on the key PK parameters of a single oral dose of midazolam in healthy postmenopausal female participants.
Part B: Area under concentration-time curve from time 0 to infinity (AUCinf) of camizestrant | Period 1 (Day 1 to Day 4), Period 2 (Day 22 to Day 25)
  To determine the effect of repeated oral titrated doses of carbamazepine on the PK of a single oral dose of camizestrant in healthy postmenopausal female participants.
Part B: Area under concentrationcurve from time 0 to the last quantifiable concentration (AUClast) of camizestrant | Period 1 (Day 1 to Day 4), Period 2 (Day 22 to Day 25)
  To determine the effect of repeated oral titrated doses of carbamazepine on the PK of a single oral dose of camizestrant in healthy postmenopausal female participants.
Part B: Maximum observed plasma (peak) drug concentration (Cmax) of camizestrant | Period 1 (Day 1 to Day 4), Period 2 (Day 22 to Day 25)
  To determine the effect of repeated oral titrated doses of carbamazepine on the PK of a single oral dose of camizestrant in healthy postmenopausal female participants.

SECONDARY OUTCOMES:
Part A: Time to reach maximum observed concentration (tmax) of midazolam | Period 1 (Day 1) and Period 3 (Day 7 to Day 8)
  To further characterise the effect of camizestrant on the PK of midazolam, and the effect of carbamazepine on the PK of camizestrant, in healthy post-menopausal female participants.
Part A: Terminal elimination half-life (t½λz) of midazolam | Period 1 (Day 1) and Period 3 (Day 7 to Day 8)
  To further characterise the effect of camizestrant on the PK of midazolam, and the effect of carbamazepine on the PK of camizestrant, in healthy post-menopausal female participants.
Part A: Terminal rate constant (λz) of midazolam | Period 1 (Day 1) and Period 3 (Day 7 to Day 8)
  To further characterise the effect of camizestrant on the PK of midazolam, and the effect of carbamazepine on the PK of camizestrant, in healthy post-menopausal female participants.
Part A: Apparent total body clearance (CL/F) of midazolam | Period 1 (Day 1) and Period 3 (Day 7 to Day 8)
  To further characterise the effect of camizestrant on the PK of midazolam, and the effect of carbamazepine on the PK of camizestrant, in healthy post-menopausal female participants.
Part A: Apparent volume of distribution based on the terminal phase (Vz/F) of midazolam | Period 1 (Day 1) and Period 3 (Day 7 to Day 8)
  To further characterise the effect of camizestrant on the PK of midazolam, and the effect of carbamazepine on the PK of camizestrant, in healthy post-menopausal female participants.
Part A: Plasma concentration of camizestrant | Period 3: Pre-dose and 3 hours post-dose of Day 7 and Day 8
  To further characterise the effect of camizestrant on the PK of midazolam, and the effect of carbamazepine on the PK of camizestrant, in healthy post-menopausal female participants.
Part B: Time to reach maximum observed concentration (tmax) of camizestrant | Period 1 (Day 1 to Day 4), Period 2 (Day 22 to Day 25)
  To further characterise the effect of camizestrant on the PK of midazolam, and the effect of carbamazepine on the PK of camizestrant, in healthy post-menopausal female participants.
Part B: Terminal elimination half-life (t½λz) of camizestrant | Period 1 (Day 1 to Day 4), Period 2 (Day 22 to Day 25)
  To further characterise the effect of camizestrant on the PK of midazolam, and the effect of carbamazepine on the PK of camizestrant, in healthy post-menopausal female participants.
Part B: Terminal rate constant (λz) of camizestrant | Period 1 (Day 1 to Day 4), Period 2 (Day 22 to Day 25)
  To further characterise the effect of camizestrant on the PK of midazolam, and the effect of carbamazepine on the PK of camizestrant, in healthy post-menopausal female participants.
Part B: Apparent total body clearance (CL/F) of camizestrant | Period 1 (Day 1 to Day 4), Period 2 (Day 22 to Day 25)
  To further characterise the effect of camizestrant on the PK of midazolam, and the effect of carbamazepine on the PK of camizestrant, in healthy post-menopausal female participants.
Part B: Apparent volume of distribution based on the terminal phase (Vz/F) of camizestrant | Period 1 (Day 1 to Day 4), Period 2 (Day 22 to Day 25)
  To further characterise the effect of camizestrant on the PK of midazolam, and the effect of carbamazepine on the PK of camizestrant, in healthy post-menopausal female participants.
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | For SAEs - Part A: From screening (Day -28 to Day -2) to 7 weeks; Part B: From screening (Day -28 to Day -2) to 9 weeks. For AEs: Part A: From Day 1 to 7 weeks; Part B: From Day 1 to 9 weeks
  To evaluate the safety and tolerability of camizestrant, alone and in combination with midazolam and carbamazepine, respectively, in healthy post-menopausal female participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/